CLINICAL TRIAL: NCT02412735
Title: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of a Single Injection of Rexlemestrocel-L Alone or Combined With Hyaluronic Acid (HA) in Subjects With Chronic Low Back Pain
Brief Title: Placebo-controlled Study to Evaluate Rexlemestrocel-L Alone or Combined With Hyaluronic Acid in Participants With Chronic Low Back Pain
Acronym: MSB-DR003
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSB-DR003
Record Dates: First submitted 2015-03-25; First posted 2015-04-09 (Estimated); Results first posted 2022-01-18 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-09

CONDITIONS: Degenerative Disc Disease
Keywords: Chronic Lumbar Back Pain; Low back pain; Back pain; Degenerative Disc Disease; Injection of Degenerated Lumbar Disc; Intervertebral Disc Degeneration; Bone Diseases; Musculoskeletal Diseases; Nervous System Diseases; Neurologic Manifestations; Pain; Spinal Diseases; Stem Cells; Adult Stem Cells; Allogeneic Mesenchymal Precursor cells (MPCs); Mesoblast; Hyaluronic Acid; Pharmaceutical Solutions; Adjuvants, Immunologic; Immunologic Factors; Pharmacologic Actions; Protective Agents; rexlemestrocel-L; Viscosupplements
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain; Back Pain; Bone Diseases; Musculoskeletal Diseases; Nervous System Diseases; Neurologic Manifestations; Pain; Spinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rexlemestrocel-L (Experimental): Participants received rexlemestrocel-L 2.0 mL injection of approximately 6 million rexlemestrocel-L cells in freeze media mixed in a 1:1 by-volume ratio with saline on Day 0 (Visit 2).
  Interventions: Drug: Rexlemestrocel-L
- Rexlemestrocel-L + HA (Experimental): Participants received rexlemestrocel-L 2.0 mL injection of approximately 6 million rexlemestrocel-L cells in freeze media mixed in a 1:1 by-volume ratio with hyaluronic acid (HA) solution on Day 0 (Visit 2).
  Interventions: Drug: Rexlemestrocel-L + HA Mixture
- Placebo (Placebo Comparator): Participants received saline solution as matching-placebo on Day 0 (Visit 2).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rexlemestrocel-L — Rexlemestrocel-L injection
  Arms: Rexlemestrocel-L
Drug: Rexlemestrocel-L + HA Mixture — Rexlemestrocel-L was combined in 1:1 by-volume ratio with HA solution and the resulting mixture was injected
  Arms: Rexlemestrocel-L + HA
Drug: Placebo — Saline control solution
  Arms: Placebo

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled Phase 3 study designed to evaluate the safety and efficacy of Mesoblast's rexlemestrocel-L alone or combined with hyaluronic acid (HA) in participants with chronic low back pain (> 6 months) associated with moderate radiographic degenerative changes of a disc.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 years of age and older
* If female of childbearing potential, participant is non-pregnant, non-nursing, and agrees to use highly effective methods of contraception for a minimum of 24 months post-treatment
* Signed informed consent and country-appropriate privacy forms indicating participant is willing to undergo treatment and willing to be available for each examination scheduled over the study duration
* Have documented diagnosis of moderate radiographic degeneration of an intervertebral disc from L1 to S1, with a disc suspected of causing chronic low back pain (CLBP) associated with moderate radiographic degeneration at a lumbar disc is defined as the following (participant must meet all of the listed conditions):

  1. Chronic low back pain for at least 6 months
  2. Have failed 6 months of conservative back pain care. (Conservative treatment regimens may include any or all of the following: initial rest, medications [e.g., anti-inflammatory, analgesics, narcotics/opioids, muscle relaxants], massage, acupuncture, chiropractic manipulations, activity modification, home-directed lumbar exercise program, and non-invasive pain control treatments or procedures)
  3. Have at a minimum undergone supervised physical therapy, such as daily walking routines, therapeutic exercises, and back education programs specifically for the treatment of low back pain and taken a pain medication for back pain (e.g. non-steroidal anti-inflammatory drug (NSAID) and/or opioid medication).
  4. Change from normal disc morphology of the index disc as defined by radiographic evaluation by the core imaging evaluation provider. Radiographs must show all of the following:
* A modified Pfirrmann score of 3, 4, 5 or 6 on magnetic resonance imaging (MRI) at the index disc
* Modic Grade II changes or less on MRI at the index disc
* With or without contained disc protrusion at the index disc on MRI

  e. Low back pain of at least 40mm and not more than 90mm of 100mm on low back pain visual analogue scale (VAS) (average pain over 24 hours)

  f. Leg pain ≤20mm in both legs on a 100mm VAS scale

  g. Oswestry disability index (ODI) score of at least 30 and no more than 90 on a 100 point scale.

Exclusion Criteria:

* Female participants who are pregnant or nursing, or women planning to become pregnant in the first 24 months post-treatment
* Extreme obesity, as defined by National Institutes of Health (NIH) Clinical Guidelines Body Mass Index (BMI > 40)
* Have undergone a surgical procedure (e.g. discectomy, intradiscal electrothermal therapy, intradiscal radiofrequency, artificial disc replacement, interbody fusion) on the disc at the index or adjacent level
* Osteoporosis, as defined by dual-energy X-ray absorptiometry (DEXA) scan. A DEXA T-score of ≤ -2.5 will exclude the participant.
* Any lumbar intradiscal injection, including steroids, into the index or adjacent discs prior to treatment injection, with the exception of the following injections performed at least 2 weeks prior to study treatment:

  1. Contrast medium (discography or other diagnostic injection)
  2. NSAIDs
  3. Nerve-blocking anesthetics (e.g., lidocaine, bupivacaine)
  4. Antibiotics
  5. Saline
* Have undergone a procedure affecting the structure/biomechanics of the index disc level (e.g., posterolateral fusion)
* Active malignancy or tumor as source of symptoms or history of malignancy within the 5 years prior to enrolment on study
* Have been a recipient of prior allogeneic stem cell/progenitor cell therapy for any indication or autologous stem cell/progenitor cell therapy or other biological intervention to repair the index intervertebral disc
* An average baseline morphine equivalent dose (MED) of >75mg/day as determined by e-diary entries during the screening period
* Taking systemic immunosuppressants
* A medical condition, serious intercurrent illness, or extenuating circumstance that would preclude participation in the study or potentially decrease survival or interfere with ambulation or rehabilitation.
* Participants involved in spinal litigation, including workman's compensation, unless litigation is complete
* Are transient or has a severe alcohol or substance abuse problem
* Clinically significant nerve pain (e.g., chronic radiculopathy or neuropathy)
* Clinically significant sacroiliac joint pain
* Compressive pathology due to stenosis or disc protrusion on MRI with associated clinical symptoms defined as leg pain VAS>20mm out of 100mm or neurologic deficit on neurologic exam
* Disc extrusion with a maximum dimension greater or equal to twice the posterior height of the disc, or disc sequestration in the lumbar spine on MRI as determined by radiographic core lab
* Modified Pfirrmann score of 7 or 8 at any lumbar level (L1-S1) on MRI evaluation as determined by radiographic core lab
* Symptomatic involvement of more than one lumbar disc
* Symptomatic central vertebral canal stenosis as defined by neurogenic claudication
* Spondylolisthesis or retrolisthesis Grade 2 and above or Spondylolysis at the index or adjacent level(s)
* Lumbar spondylitis or other undifferentiated spondyloarthropathy affecting the index disc
* Spinal deformity defined as lumbar scoliosis with a Cobb angle of the lumbar spine greater than 15 degrees
* Any fracture of the spine at the index or adjacent levels that has not healed, or clinically compromised vertebral bodies at the index level due to current or past trauma
* Facet pain at the index level or adjacent segments as determined by a diagnostic medial branch block (a facet block injection is not acceptable for making this determination) to rule out facet joint involvement.
* Full thickness annular tears in the index level as determined by free flowing contrast media through the annulus fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brown, Study Director — Mesoblast, Ltd.
Locations (48):
- United States (47):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Tennessee Valley Pain Consultants, Huntsville, Alabama
  - Arizona Pain Specialists, Scottsdale, Arizona
  - Physicians Research Group, Tempe, Arizona
  - TriWest Research Associates, LLC, El Cajon, California
  - Memorial Orthopaedics Surgical Group, Long Beach, California
  - Newport Beach Headache and Pain, Newport Beach, California
  - Institute for Regenerative Medicine and Clinical Research, Pasadena, California
  - UC Davis Spine Center, Sacramento, California
  - Orthopedic Pain Specialists, Santa Monica, California
  - The Spine Institute, Santa Monica, California
  - Summit Pain Alliance, Santa Rosa, California
  - Integrated Pain Management, Walnut Creek, California
  - Denver Back Pain Specialists, LLC, Greenwood Village, Colorado
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Coastal Clinical Research Specialists, Fernandina Beach, Florida
  - Shrock Orthopedic Research, LLC, Fort Lauderdale, Florida
  - Holy Cross Orthopedics Institute, Oakland Park, Florida
  - Emory Orthopaedics & Spine Center, Atlanta, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Injury Care Medical Center, Boise, Idaho
  - Millennium Pain Center, Bloomington, Illinois
  - Otrimed Clinical Research, Edgewood, Kentucky
  - Orthopedic Specialists of Louisiana, Shreveport, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - MAPS Applied Research Center, Shakopee, Minnesota
  - Innovative Pain Care Center, Las Vegas, Nevada
  - University Clinical Research, Somerset, New Jersey
  - Ainsworth Institute of Pain Management, New York, New York
  - Rochester Regional Health, Rochester, New York
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - On Site Clinical Solutions, LLC, Morrisville, North Carolina
  - The Center for Clinical Research/ Carolinas Pain Institute, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - DOC Clinical Research, Dayton, Ohio
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - Orthopaedic and Spine Specialists, York, Pennsylvania
  - RI Hospital-Comprehensive Spine Center, Providence, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Greenville Pharmaceutical Research, Inc., Charleston, South Carolina
  - Texas Back Institute, Plano, Texas
  - Spine Team Texas, Southlake, Texas
  - Precision Spine Care, Tyler, Texas
  - Ericksen Research & Development, LLC, Bountiful, Utah
  - the SMART Clinic, Draper, Utah
  - Hope Research Institute, St. George, Utah
  - Virginia iSpine Physicians, PC, Richmond, Virginia
- Monash Medical Center, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Starting on March 6, 2015, a total of 404 participants were enrolled at investigative sites in Australia and the United States.
Period: Overall Study
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
Started | 143 | 129 | 132
Received Treatment | 140 | 128 | 130
Completed | 97 | 85 | 86
Not Completed | 46 | 44 | 46
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Withdrawal by Subject | 23 | 27 | 22
Not completed — Investigator Decision | 3 | 3 | 2
Not completed — Lost to Follow-up | 17 | 11 | 18
Not completed — Reason not Specified | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) Analysis Set included all participants who were randomized, regardless of whether or not the participant was treated, or post-treatment measures were performed.
Groups:
- Rexlemestrocel-L + HA: Participants received rexlemestrocel-L 2.0 mL injection of approximately 6 million rexlemestrocel-L cells in freeze media mixed in a 1:1 by-volume ratio with HA solution on Day 0 (Visit 2).
- Total: Total of all reporting groups
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo | Total
Number analyzed (Participants) | 143 | 129 | 132 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (10.81) | 42.9 (11.66) | 43.3 (10.45) | 42.8 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 54 | 61 | 175
  Male | 83 | 75 | 71 | 229
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 11 | 24
  Not Hispanic or Latino | 133 | 121 | 119 | 373
  Unknown or Not Reported | 1 | 4 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 6 | 18
  White | 133 | 118 | 118 | 369
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Treatment Success: Bayesian Estimated Response Rate
Description: Overall treatment success was determined based on number of responders who had composite response at both months 12 and 24 evaluated per specified criteria. A treatment responder with treatment success was defined as a participant who met the 3 criteria of a composite responder analysis as: 50% or greater reduction in the lower-back pain visual analogue scale (VAS) score; 15-point or greater reduction in the Oswestry Disability Index (ODI) score; and lack of post-treatment interventions at the treated level as of the study visit (Visits 6 [12 months post-treatment] and 8 [24 months post-treatment]). The average response rate (proportion of participants with response presented as Bayesian estimate[BE]) was based upon the average of multiple Bayesian simulations.
Time Frame: Up to 24 months
Population: The ITT Analysis Set included all participants who were randomized, regardless of whether or not the participant was treated, or post-treatment measures were performed.
Measure: Mean (Standard Deviation); unit: BE proportion of participants
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
Number analyzed (Participants) | 143 | 129 | 132
BE proportion of participants | 0.267 (0.038) | 0.335 (0.043) | 0.313 (0.041)
Statistical Analysis 1: Comparison: Rexlemestrocel-L vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.2072
Statistical Analysis 2: Comparison: Rexlemestrocel-L + HA vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.6427

2. Secondary Outcome: Effectiveness Based on Pain Responders: Bayesian Estimated Response Rate
Description: A participant was defined as a pain responder for a given study visit if they achieved at least a 50% reduction from Baseline in the lower-back pain VAS score (average pain over 24 hours), as reported during in-clinic assessment. The participant should be qualified as a pain responder at both 12 and 24 months post-treatment, and must not have received a post-treatment intervention through 24 months' follow-up. Any participant that did not have a minimum of a visit at 3 months (Study Visit 4) was considered a non-responder for this outcome measure. The average response rate (proportion of participants with response presented as BE) was based upon the average of multiple Bayesian simulations.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BE proportion of participants
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
Number analyzed (Participants) | 143 | 129 | 132
BE proportion of participants | 0.352 (0.041) | 0.472 (0.045) | 0.388 (0.044)
Statistical Analysis 1: Comparison: Rexlemestrocel-L vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.2754
Statistical Analysis 2: Comparison: Rexlemestrocel-L + HA vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.9087

3. Secondary Outcome: Effectiveness Based on Functional Responders: Bayesian Estimated Response Rate
Description: A participant was defined as a functional responder for a given study visit if they achieved at least a 15-point reduction from Baseline in ODI score, as reported during in-clinic assessment. The participant should be qualified as a functional responder at both 12 and 24 months post-treatment, and must not have received a post-treatment intervention through 24 months' follow-up; any participant that did not have a minimum of a visit at 3 months (Study Visit 4) was considered a non-responder for this outcome measure. The average response rate (proportion of participants with response presented as BE) was based upon the average of multiple Bayesian simulations.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BE proportion of participants
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
Number analyzed (Participants) | 143 | 129 | 132
BE proportion of participants | 0.378 (0.042) | 0.409 (0.045) | 0.413 (0.044)
Statistical Analysis 1: Comparison: Rexlemestrocel-L vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.2835
Statistical Analysis 2: Comparison: Rexlemestrocel-L + HA vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.4739

4. Secondary Outcome: Effectiveness Based on Treatment Success at 24 Months: Bayesian Estimated Response Rate
Description: A treatment responder with treatment success was defined as a participant who met the 3 conditions of a composite responder analysis as: 50% or greater reduction in the lower-back pain VAS score; 15-point or greater reduction in ODI score; and lack of post-treatment interventions at the treated level as of the study visit. The participants qualified as responders if they satisfied the above conditions at the 24-month follow-up visit alone. Any participant that did not have a minimum of a visit at 3 months (Study Visit 4) was considered a non-responder for this outcome measure. The average response rate (proportion of participants with response presented as BE) was based upon the average of multiple Bayesian simulations.
Time Frame: Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BE proportion of participants
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
Number analyzed (Participants) | 143 | 129 | 132
BE proportion of participants | 0.353 (0.042) | 0.425 (0.045) | 0.391 (0.045)
Statistical Analysis 1: Comparison: Rexlemestrocel-L vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.2650
Statistical Analysis 2: Comparison: Rexlemestrocel-L + HA vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.7004

5. Secondary Outcome: Effectiveness Based on Minimal Pain Responders at 24 Months: Bayesian Estimated Response Rate
Description: A minimal pain responder was defined as a participant who achieved a lower-back pain VAS score (average pain over 24 hours) of 20 mm or less at the given study visit. The participants qualified as responders if they satisfied the above condition at 24 months post-treatment, and did not receive a post-treatment intervention through 24 months' follow-up. Any participant that did not have a minimum of a visit at 3 months (Study Visit 4) was considered a non-responder for this outcome measure. The average response rate (proportion of participants with response presented as BE) was based upon the average of multiple Bayesian simulations.
Time Frame: Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BE proportion of participants
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
Number analyzed (Participants) | 143 | 129 | 132
BE proportion of participants | 0.384 (0.043) | 0.495 (0.047) | 0.438 (0.046)
Statistical Analysis 1: Comparison: Rexlemestrocel-L vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.1945
Statistical Analysis 2: Comparison: Rexlemestrocel-L + HA vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.8093

6. Secondary Outcome: Effectiveness Based on Time to First Intervention Over 24 Months
Description: The effectiveness of the study drug was evaluated based on its ability in increasing the time to additional interventions at the treated level over 24 months post-treatment. Kaplan-Meier estimates for the probability (expressed as a percentage) of participants to receive an intervention are presented.
Time Frame: Up to Month 24
Population: as for outcome 1
Measure: Number; unit: percentage probability
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
Number analyzed (Participants) | 143 | 129 | 132
percentage probability | 0.1099 | 0.1003 | 0.0913
Statistical Analysis 1: Comparison: Rexlemestrocel-L vs Placebo; Test type: Superiority; p = 0.7842, Regression, Cox; P-value was calculated from a Cox regression model with treatment, pooled site, and opioid/non opioid use at Baseline as covariates; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.50 to 2.46] — Hazard ratio and 95% confidence interval (CI) were calculated from a Cox regression model with treatment, pooled site, and opioid/non opioid use at Baseline as covariates
Statistical Analysis 2: Comparison: Rexlemestrocel-L + HA vs Placebo; Test type: Superiority; p = 0.8754, Regression, Cox; [statistical method as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.41 to 2.14] — Hazard ratio and 95% CI were calculated from a Cox regression model with treatment, pooled site, and opioid/non opioid use at Baseline as covariates

7. Secondary Outcome: Effectiveness Based on Minimal Disability Responders at 24 Months: Bayesian Estimated Response Rate
Description: A minimal disability responder was defined as a participant who achieved an ODI score of 20% or less at the given study visit. The participants qualified as responders if they satisfied the above condition at 24 months post-treatment, and did not receive a post-treatment intervention through 24 months' follow-up. Any participant that did not have a minimum of a visit at 3 months (Study Visit 4) was considered a non-responder for this outcome measure. The average response rate (proportion of participants with response presented as BE) was based upon the average of multiple Bayesian simulations.
Time Frame: Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BE proportion of participants
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
Number analyzed (Participants) | 143 | 129 | 132
BE proportion of participants | 0.394 (0.043) | 0.367 (0.045) | 0.440 (0.045)
Statistical Analysis 1: Comparison: Rexlemestrocel-L vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.2309
Statistical Analysis 2: Comparison: Rexlemestrocel-L + HA vs Placebo; Test type: Superiority — The superiority threshold was 0.9875; The posterior probability of superiority to placebo was 0.1241

8. Other Pre Specified Outcome: Mean Change From Baseline in Low Back Pain Visual Analog Scale (VAS) Score at 1, 3, 6, 12, 18, 24, and 36 Months
Description: Pain intensity was recorded on a horizontal 100 mm VAS and measured as the distance in millimeters from the left origin of the horizontal VAS line and the point indicated by the participant as representing their level of pain. A horizontal 100 mm VAS anchored on the left with the words "No Pain" and on the right with the words "Worst Possible Pain", was used to measure low back pain intensity. Scores were obtained by measuring the distance in millimeters from the left origin of the line (0) to the point indicated with a slash placed by the participant to indicate the participant's level of pain. VAS ranges from 0 to 100, with higher scores indicating worst possible pain. A negative change from baseline indicates improvement.
Time Frame: Months 1, 3, 6, 12, 18, 24, and 36
Population: The ITT Analysis Set included all participants who were randomized, regardless of whether or not the participant was treated, or post-treatment measures were performed. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
Number analyzed (Participants) | 143 | 129 | 132
score on a scale
  Change from Baseline at Month 1: number analyzed (Participants) | 139 | 125 | 124
  Change from Baseline at Month 1 | -13.6 (2.14) | -17.3 (2.30) | -13.9 (2.32)
  Change from Baseline at Month 3: number analyzed (Participants) | 130 | 120 | 124
  Change from Baseline at Month 3 | -19.1 (2.26) | -22.5 (2.41) | -17.6 (2.40)
  Change from Baseline at Month 6: number analyzed (Participants) | 129 | 116 | 124
  Change from Baseline at Month 6 | -22.4 (2.34) | -24.9 (2.51) | -18.6 (2.48)
  Change from Baseline at Month 12: number analyzed (Participants) | 121 | 111 | 117
  Change from Baseline at Month 12 | -23.3 (2.38) | -27.4 (2.55) | -19.0 (2.51)
  Change from Baseline at Month 18: number analyzed (Participants) | 110 | 99 | 104
  Change from Baseline at Month 18 | -23.7 (2.56) | -25.1 (2.74) | -19.2 (2.70)
  Change from Baseline at Month 24: number analyzed (Participants) | 112 | 99 | 102
  Change from Baseline at Month 24 | -20.8 (2.55) | -25.9 (2.74) | -18.3 (2.70)
  Change from Baseline at Month 36: number analyzed (Participants) | 99 | 89 | 90
  Change from Baseline at Month 36 | -22.9 (2.62) | -25.1 (2.81) | -19.0 (2.77)
Statistical Analysis 1: Comparison: Rexlemestrocel-L vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 1; Test type: Superiority; p = 0.9072, Mixed Model for Repeated Measures (MMRM); MMRM was used with fixed effects of pooled site,baseline use of opioids,treatment,visit,treatment-by-visit interaction&continuous covariate baseline; Least Squares Mean Difference = 0.4, 95% CI 2-sided [-5.71 to 6.43], Standard Error of Mean 3.08
Statistical Analysis 2: Comparison: Rexlemestrocel-L + HA vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 1; Test type: Superiority; p = 0.2883, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -3.3, 95% CI 2-sided [-9.51 to 2.83], Standard Error of Mean 3.14
Statistical Analysis 3: Comparison: Rexlemestrocel-L vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 3; Test type: Superiority; p = 0.6314, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -1.6, 95% CI 2-sided [-7.90 to 4.80], Standard Error of Mean 3.23
Statistical Analysis 4: Comparison: Rexlemestrocel-L + HA vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 3; Test type: Superiority; p = 0.1366, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -4.9, 95% CI 2-sided [-11.37 to 1.56], Standard Error of Mean 3.29
Statistical Analysis 5: Comparison: Rexlemestrocel-L vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 6; Test type: Superiority; p = 0.2497, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -3.9, 95% CI 2-sided [-10.43 to 2.72], Standard Error of Mean 3.34
Statistical Analysis 6: Comparison: Rexlemestrocel-L + HA vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 6; Test type: Superiority; p = 0.0666, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -6.3, 95% CI 2-sided [-13.00 to 0.43], Standard Error of Mean 3.42
Statistical Analysis 7: Comparison: Rexlemestrocel-L vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 12; Test type: Superiority; p = 0.2147, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -4.2, 95% CI 2-sided [-10.91 to 2.46], Standard Error of Mean 3.40
Statistical Analysis 8: Comparison: Rexlemestrocel-L + HA vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 12; Test type: Superiority; p = 0.0162, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -8.4, 95% CI 2-sided [-15.19 to -1.55], Standard Error of Mean 3.47
Statistical Analysis 9: Comparison: Rexlemestrocel-L vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 18; Test type: Superiority; p = 0.2230, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -4.5, 95% CI 2-sided [-11.69 to 2.74], Standard Error of Mean 3.67
Statistical Analysis 10: Comparison: Rexlemestrocel-L + HA vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 18; Test type: Superiority; p = 0.1152, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -5.9, 95% CI 2-sided [-13.27 to 1.45], Standard Error of Mean 3.74
Statistical Analysis 11: Comparison: Rexlemestrocel-L vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 24; Test type: Superiority; p = 0.4884, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -2.5, 95% CI 2-sided [-9.75 to 4.67], Standard Error of Mean 3.66
Statistical Analysis 12: Comparison: Rexlemestrocel-L + HA vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 24; Test type: Superiority; p = 0.0426, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -7.6, 95% CI 2-sided [-14.98 to -0.25], Standard Error of Mean 3.74
Statistical Analysis 13: Comparison: Rexlemestrocel-L vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 36; Test type: Superiority; p = 0.3056, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -3.9, 95% CI 2-sided [-11.27 to 3.54], Standard Error of Mean 3.77
Statistical Analysis 14: Comparison: Rexlemestrocel-L + HA vs Placebo; Mean Change from Baseline in Low Back Pain VAS Score at Month 36; Test type: Superiority; p = 0.1184, MMRM; [statistical method as in outcome 8, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-13.59 to 1.54], Standard Error of Mean 3.85

ADVERSE EVENTS:
Time Frame: Up to approximately 38 months
Description: All-cause Mortality: The ITT Analysis Set included all participants who were randomized, regardless of whether or not the participant was treated, or post-treatment measures were performed. Serious and Other (Non-serious) Adverse Events: Safety Analysis Set included all participants who were randomized and received treatment, and classified according to the actual treatment received.
Arm/Group | Rexlemestrocel-L | Rexlemestrocel-L + HA | Placebo
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/129 | 0/132
Serious Adverse Events (participants affected / at risk) | 17/140 | 15/128 | 10/130
Other Adverse Events (participants affected / at risk) | 111/140 | 100/128 | 98/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rexlemestrocel-L (N=140) | Rexlemestrocel-L + HA (N=128) | Placebo (N=130)
Appendicitis (Infections and infestations) | 2 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Escherichia bacteremia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Perineurial cyst (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Sacral radiculopathy (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Spinal meningeal cyst (Nervous system disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic hematoma (Hepatobiliary disorders) | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Device breakage (Product Issues) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Investigations (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Influenza b virus test positive (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hip surgery (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rexlemestrocel-L (N=140) | Rexlemestrocel-L + HA (N=128) | Placebo (N=130)
Back pain (Musculoskeletal and connective tissue disorders) | 51 | 56 | 48
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 17 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 15 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 7 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 10
Hypoesthesia (Nervous system disorders) | 10 | 8 | 12
Paresthesia (Nervous system disorders) | 11 | 5 | 4
Nausea (Gastrointestinal disorders) | 5 | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications (abstracts, posters or presentations) must be presented to the Publication Steering Committee for review prior to submission or public display and are not allowed prior to the publication of the primary manuscript, or eighteen (18) months from the conclusion of the Study. PI shall provide Sponsor a copy of any proposed public disclosure at least 30 days prior to submission. Sponsor may ask PI to delay the disclosure for a maximum of 60 days to file proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT02412735/Prot_SAP_001.pdf